CLINICAL TRIAL: NCT03674736
Title: Application of the Indicator Amino Acid Oxidation Technique for the Determination of Metabolic Availability of Methionine and Lysine From Rice, Wheat, Chickpeas and Lentils, in Healthy Young Adult Men
Brief Title: Metabolic Availability of Methionine and Lysine From Rice, Wheat, Chickpea and Lentil in Adult Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Project Investigator, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000061263
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Healthy; Men; Adults; Methionine; Lysine
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Eating

STUDY DESIGN:
Intervention Model Description: Each subject will randomly receive 4 levels of methionine or lysine provided as free amino acids, Rice, Wheat, Chickpeas or Lentils for a total of 7 studies x 3 days per study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Methionine bioavailability in Rice (Experimental): Participants will be seen initially for pre-study assessment (3 hour). They will then be studied for up to 7 times. You could be expected to participate in up to 7 different sets of experiments which will take 8 weeks to 6 months. Each set of experiment consists of a 3 day period. During the first 2 days (Adaptation Days) you will be expected to consume 4 meals per day consisting of a protein liquid drink and protein freecookies and/or Rice which will be provided by the investigators
  Interventions: Dietary Supplement: Dietary Intakes
- Lysine bioavailability in Chickpeas (Experimental): Participants will be seen initially for pre-study assessment (3 hour). They will then be studied for up to 7 times. You could be expected to participate in up to 7 different sets of experiments which will take 8 weeks to 6 months. Each set of experiment consists of a 3 day period. During the first 2 days (Adaptation Days) you will be expected to consume 4 meals per day consisting of a protein liquid drink and protein freecookies and/or Chickpeas which will be provided by the investigators
  Interventions: Dietary Supplement: Dietary Intakes
- Methionine bioavailability in Wheat (Experimental): Participants will be seen initially for pre-study assessment (3 hour). They will then be studied for up to 7 times. You could be expected to participate in up to 7 different sets of experiments which will take 8 weeks to 6 months. Each set of experiment consists of a 3 day period. During the first 2 days (Adaptation Days) you will be expected to consume 4 meals per day consisting of a protein liquid drink and protein freecookies and/or Wheat bread which will be provided by the investigators
  Interventions: Dietary Supplement: Dietary Intakes
- Lysine bioavailability in Lentils (Experimental): Participants will be seen initially for pre-study assessment (3 hour). They will then be studied for up to 7 times. You could be expected to participate in up to 7 different sets of experiments which will take 8 weeks to 6 months. Each set of experiment consists of a 3 day period. During the first 2 days (Adaptation Days) you will be expected to consume 4 meals per day consisting of a protein liquid drink and protein freecookies and/or Lentils which will be provided by the investigators
  Interventions: Dietary Supplement: Dietary Intakes

INTERVENTIONS:
Dietary Supplement: Dietary Intakes — Four levels of methionine or lysine intakes will be provided by the reference protein drinks, 3 levels of methionine from rice and wheat bread and 3 levels of lysine from chickpeas and lentils

SUMMARY:
The research study is being done so we can determine the quality of the protein present in Rice, Wheat, Chickpeas and Lentils. Amino acids are the building blocks of protein and protein quality is determined by the amount of amino acids present and by their bioavailability (their absorption and use by the body). Some amino acids are essential which means they must be obtained from the diet. If any one of the essential amino acids is missing in the diet, the body cannot make proteins that are used to repair tissue build bone, teeth, etc… Rice, Wheat, Chickpeas and Lentils as a food source contain low amounts of the essential amino acid methionine (Chickpeas and Lentils) and lysine (Rice and Wheat) which makes its protein incomplete. The amino acids in Rice, Wheat, Chickpeas and Lentils are also affected by cooking. Our objective is to determine the amount of methionine in Rice and Wheat and the amount of lysine in Chickpeas and Lentils that the body can use.

This research is being done in order to bridge the gap between knowledge of protein requirement and the amount of food needed to meet that requirement. Results from this study will be important for recommendations guiding food choices of Rice, Wheat, Chickpeas and Lentils as a major protein source in the diet.

Previously the quality of dietary protein for human consumption was studied in animals. This study is being done in humans because studies in animals are not always directly applicable to humans. Plant protein sources like rice, wheat, chickpeas and lentils are important protein sources shown to "enhance ecosystem resilience, and improve human health.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will participate in 7 different experiments for each food. For each food you will receive 3 different amounts of Rice, Wheat, Chickpeas or Lentils which will contain different amounts of the essential amino acid methionine (Rice or Wheat) or lysine (Chickpeas or Lentils).

The quality of the protein in the Rice, Wheat, Chickpeas or Lentils will be compared to the quality of a reference protein (egg protein) by giving you 4 reference diets containing amino acids made up like the amino acids in egg protein. The amount of Rice, Wheat, Chickpeas or Lentils you receive will be provided in a random order.

Each experiments will be conduced over 3 days- 2 adaptation days where you will receive the diets at home, provided by the investigators and 1 study day. On the 3rd day (study day) you will visit the Clinical Research Center (CRC) at the Hospital for Sick Children where you will receive 9 hourly meals. Breath samples will be collected after the 4th meal in 15 min intervals for 1 hour. Breath collection will resume again two and a half hours after the 5th meal every 15 minutes until 30 minutes after the last meal. A total of 52 breath samples will be collected during each of the 3rd study day.

Before the study begins, you will visit the CRC at the Hospital for Sick Children for a baseline study assessment. At that time your body composition (fat and fat-free mass) will be measured and your resting energy expenditure will be measured. This will tell us the amount of calories your body need so we can prepare the diets for you for each experiment. This baseline assessment takes about 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18 - 49 yrs, Healthy with no known clinical condition which would affect protein or AA metabolism, ex. Diabetes, Stable Body Weight (no more than 5 lb weight loss or gain in the past 3 months) Not on any medications that could affect protein or amino acid metabolism e.g. steroids

Exclusion Criteria:

* Unwillingness to participate or unable to tolerate the diet Recent history of weight loss within the last 3 months or on a weight reducing diet Inability to tolerate study diets (ex. Allergy to ingredients).

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Metabolic availability of Methionine in Rice Apply the IAAO method to determine the MA of methionine in Canadian grown lentils prepared by moist cooking method. | 2 years
  Apply the IAAO method to determine the MA of methionine in rice method.
Metabolic availability of Methionine in Wheat | 2 years
  Apply the IAAO method to determine the MA of methionine in wheat bread
Metabolic availability of Lysine in Chickpeas | 2 years
  Apply the IAAO method to determine the MA of lysine in chickpeas
Metabolic availability of Lysine in Lentils | 2 years
  Apply the IAAO method to determine the MA of lysine in Canadian grown lentils

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tul-Noor Z, Paoletti A, Fakiha A, Pencharz PB, Levesque CL, Ball RO, Elango R, Courtney-Martin G. Lysine from Whole Wheat Bread Consumed by Healthy Adult Males Has High Metabolic Availability When Assessed Using the Indicator Amino Acid Oxidation Method. J Nutr. 2025 Feb;155(2):476-482. doi: 10.1016/j.tjnut.2024.08.011. Epub 2024 Aug 18. PMID 39163973
- [Derived] Fakiha A, Tul-Noor Z, Paoletti A, Pencharz PB, Ball RO, Levesque CL, Elango R, Courtney-Martin G. Bioavailable Lysine, Assessed in Healthy Young Men Using Indicator Amino Acid Oxidation, is Greater when Cooked Millet and Stewed Canadian Lentils are Combined. J Nutr. 2020 Oct 12;150(10):2729-2737. doi: 10.1093/jn/nxaa227. PMID 32840580
- [Derived] Rafii M, Pencharz PB, Ball RO, Tomlinson C, Elango R, Courtney-Martin G. Bioavailable Methionine Assessed Using the Indicator Amino Acid Oxidation Method Is Greater When Cooked Chickpeas and Steamed Rice Are Combined in Healthy Young Men. J Nutr. 2020 Jul 1;150(7):1834-1844. doi: 10.1093/jn/nxaa086. PMID 32271919